CLINICAL TRIAL: NCT03348982
Title: Examining the Association Between Physical Activity and Sleep Quality in Children With Autism Spectrum Disorder Using Melatonin-mediated Mechanism Model: A Randomized Controlled Trial
Brief Title: Examining the Association Between Physical Activity and Sleep Quality in Children With Autism Spectrum Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28602517
Record Dates: First submitted 2017-11-09; First posted 2017-11-21 (Actual); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Physical Activity; Sleep Apnea; Autism Spectrum Disorder
Keywords: Physical activity; Sleep; Children; Autism Spectrum Disorder; Melatonin
MeSH Terms: conditions — Motor Activity; Sleep Apnea Syndromes; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention is a 12-week jogging program consisting of 24 sessions (two sessions per week, 30 min per session) in a hall/gymnasium of each participating school.Each intervention session will be conducted in the morning by a trained research assistant assisted by student helpers. Each intervention session will be conducted in an identical format, comprising three activities: warm-up (5 min), jogging (20 min), and cool-down (5 min). In the jogging activity, participants will be asked to jog side-by-side with the research staff around an activity circuit (57m x 50m) marked with 4 red cones.
  Interventions: Behavioral: Jogging program
- Control group (No Intervention): Participants in the control group will receive no physical intervention and will be required to follow their daily routine without participating in any additional physical activity/exercise program throughout the whole study period (T1-T3).

INTERVENTIONS:
Behavioral: Jogging program — The intervention is a 12-week jogging program consisting of 24 sessions (two sessions per week, 30 min per session).
  Arms: Intervention group

SUMMARY:
This study aims to investigate whether physical activity intervention would be effective to improve sleep quality in children with ASD, and investigate how physical activity impacts on sleep in children with ASD through melatonin-mediated mechanism model. A parallel-group randomized controlled trial comparing a 12-week jogging intervention and a control group receiving standard care in 32 children with ASD will be conducted. This study will monitor the changes of four sleep parameters (sleep onset latency; sleep efficiency, wake after sleep onset and sleep duration) through objective actigraphic assessment and parental sleep logs.

DETAILED DESCRIPTION:
Sleep disturbance is commonly found in children with autism spectrum disorder (ASD) and is often accompanied with family distress. Disturbed sleep may exacerbate the core symptoms of ASD including stereotypic behaviors, social interactions, and health problems. Therefore, it is important to develop effective intervention strategies to ameliorate the sleep disturbance in children with ASD. Traditionally, behavioral interventions and supplemental melatonin medication are used to improve their sleep quality. However, poor sustainability of behavioral intervention effects and use of other medications (e.g. antidepressants and stimulants) that metabolize melatonin may degrade the effectiveness of these interventions. Alternatively, previous research supported physical activity intervention as an effective treatment on sleep disturbance for typically developing children who suffered from sleep disturbance. It is therefore natural to extend the study to examine whether such intervention is also effective in children with ASD. This study aims to investigate whether physical activity intervention would be effective to improve sleep quality in children with ASD. Moreover, how physical activity impacts on sleep in children with ASD through melatonin-mediated mechanism model will also be investigated. According to this mechanism model, it is suggested that physical activity could affect circadian rhythm through altering melatonin level. Melatonin is generally lower in ASD children than in their typically developing counterparts and supplemental melatonin medication is often used to treat the sleep disturbance in this population. This study is a parallel-group randomized controlled trial comparing a 12-week jogging intervention and a control group receiving standard care in 32 children with ASD. The changes of four sleep parameters (sleep onset latency; sleep efficiency, wake after sleep onset and sleep duration) through objective actigraphic assessment and parental sleep logs will be monitored. To measure melatonin level, all participants will be instructed to collect a 24-h urinary sample. 6-sulfatoxymelatonin, a creatinine-adjusted morning urinary melatonin and representative for melatonin level, will be measured from the collected urine sample. All the assessments will be carried out before the intervention (T1), immediately after the 12 weeks of physical activity intervention or regular treatment (T2), and 12 weeks after post-intervention (T3) for examination of sustained intervention effect. The findings of this proposed study can provide information on the mechanism pathway that physical activity impacts on sleep in children with ASD, which will contribute to the design of an effective intervention to improve sleep quality for children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* pre-puberty or early puberty as indicated by Tanner stage I or II ;
* ASD diagnosis from a physician based on Diagnostic and Statistical Manual of Mental Disorders, 5th edition, (DSM-V)[42]
* non-verbal IQ over 40
* the ability to follow instructions;
* physically able to participate in the intervention
* no additional regular participation in physical exercise other than school physical education classes for at least 6 months prior to the study
* no concurrent medication for at least 6 months before the study or any prior melatonin treatment;
* have sleep difficulties, including sleep onset insomnia and frequent and prolonged nightwaking and/or early morning awakenings reported by parents

Exclusion Criteria:

* with one or co-morbid psychiatric disorders as established by a structured interview based on DSM-V
* with other medical conditions that limit their physical activity capacities (e.g., asthma, seizure, cardiac disease);
* with a complex neurologic disorder (e.g., epilepsy, phenylketonuria, fragile X syndrome, tuberous sclerosis)

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Sleep onset latency | 12-week
  Sleep onset latency (length of time taken to fall asleep, expressed in minutes, SOL) will be objectively measured by a GT3X accelerometer.
Sleep efficiency | 12-week
  Sleep efficiency (actual sleep time divided by time in bed, expressed as a percent, SE) will be objectively measured by a GT3X accelerometer.
Wake after sleep onset | 12-week
  Wake after sleep onset (length of time they were awake after sleep onset, expressed in minutes, WASO) will be objectively measured by a GT3X accelerometer.
Sleep duration | 12-week
  sleep duration (total sleep in hours and minutes, SD) will be objectively measured by a GT3X accelerometer.
Parental-assessed sleep quality | 12-week
  Participants' sleep patterns will be logged by their parents using Children's Sleep Habits Questionnaire (CSHQ), which is a validated 45-item parent-administered questionnaire to examine sleep patterns of young children. The total score ranged from 45 to 135.
Melatonin | 12-week
  All participants will be instructed to collect a 24-h urine sample. 6-sulfatoxymelatonin, a creatinine-adjusted morning urinary melatonin and representative of melatonin level, will be measured from the sample. The weekend has been chosen to allow the participants to stay at home for sample collection. All urine samples will be collected using 24-h urine bottles containing 0.1L of 0.5M hydrochloric acid as a preservative.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tse ACY, Lee PH, Zhang J, Lai EWH. Study protocol for a randomised controlled trial examining the association between physical activity and sleep quality in children with autism spectrum disorder based on the melatonin-mediated mechanism model. BMJ Open. 2018 Apr 13;8(4):e020944. doi: 10.1136/bmjopen-2017-020944. PMID 29654045